CLINICAL TRIAL: NCT06579729
Title: Dietary Intervention for Low Free Sugars in Children With Non-alcoholic Fatty Liver Disease: a Randomized Controlled Trial
Brief Title: Dietary Intervention for Low Free Sugars in Children With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Haonan Zhou, Investigator, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018140037
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: NAFLD; Low-free Sugar Dietary; Child Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Dietary intervention for low free sugars
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Dietary intervention for low free sugars — After baseline data collection, the intervention group received a 30-60 minute educational session with a dietitian and clinicians, including a health education prescription. Interventions occurred at weeks 1, 12 and 24, with routine evaluations of disease, diet, physical activity, and adherence. Follow-ups at 48 weeks assessed NAFLD extent, dietary profile, and health knowledge for both subjects and guardians.
  Arms: Intervention group

SUMMARY:
A 48-week dietary intervention program was conducted in children aged 5-14 years with a diagnosis of NAFLD, who were randomized into a low free sugar diet group and a regular diet group. The primary objective of this study is to determine whether a low free sugar dietary intervention program improves liver function, fasting glucose, fasting insulin, lipid profile and hepatic steatosis in children with NAFLD. The effects of the intervention will be analyzed and compared at weeks 12, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 5 years old and below 14 years old;
* Guardian's consent and signing of informed consent;
* WHO growth and development curves as the reference standard, overweight is defined as BMI greater than or equal to the 85th percentile of the WHO growth curves for children, and obesity is defined as BMI greater than or equal to the 95th percentile of the WHO growth curves for children;
* Liver imaging performance meets the diagnostic criteria of diffuse fatty liver.

Exclusion Criteria:

* Age <5 years or >14 years;
* Previous history of alcohol consumption;
* Non-cooperation with the study, inability to comply with the study treatment or study visit.
* Past or active hepatitis B virus infection;
* Past or active hepatitis C virus infection;
* Chronic or acute liver failure;
* Cholestasis;
* Hepatomegaly;
* Cystic fibrosis;
* α1-antitrypsin deficiency;
* Autoimmune hepatitis;
* Tyrosinemia;
* Galactosemia or any recognized liver disease, any physical condition deemed by a physician to be unable to complete the trial. Physical Condition.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
NAFLD | At weeks 1, 12 and 24
  NAFLD was diagnosed using liver ultrasonography with a Phillip IU Elite color Doppler ultrasound after a fasting period to reduce gastrointestinal interference.
Dietary | At weeks 1, 12 and 24
  The dietary habits of the subjects were evaluated by a semi-quantitative Food Frequency Questionnaire (FFQ), which was recalled over the past month and included food items, frequency, and amount of intake. The FFQ used in this study covered 72 food items from 11 food groups and 4 frequency categories, including 'average daily, weekly, monthly intake or hardly eat'.
Physical activity level | At weeks 1, 12 and 24
  Physical Activity Questionnaire for Children (PAQ-C) was answered by subjects. The PAQ-C reflects the overall physical activity level of children in the past 7 days.The scale consists of 10 items, .and a 1-5 scale was used to obtain a total score by summing the scores of the individual items. The PAQ-C scale scores < 2.33 defined as low physical activity levels, 2.33-3.66 as moderate physical activity levels, and >3.66 as high physical activity levels.

SECONDARY OUTCOMES:
Height | At weeks 1, 12 and 24
  Height was measured using Height Measuring Ruler (Selcom, Germany) .
Body weight | At weeks 1, 12 and 24
  Body weight was measured using Body Composition Analyzer (DC-13, Parade, Japan).
BMI | At weeks 1, 12 and 24
  BMI (kg/m2) = body weight (kg)/height2 (m2).
Waist circumference | At weeks 1, 12 and 24
  Waist circumference was measured with circumference measuring tape.
Waist-to-height ratio | At weeks 1, 12 and 24
  Waist-to-height ratio (WHtR) = waist circumference (cm)/height (cm).
Blood pressure | At weeks 1, 12 and 24
  Blood pressure was measured using an Omron electronic blood pressure monitor (HBP-1300).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Shenyang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT06579729/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT06579729/ICF_001.pdf